CLINICAL TRIAL: NCT01843777
Title: Applying the Use of Motivational Tools to Auditory Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C1004-P
Record Dates: First submitted 2013-04-23; First posted 2013-05-01 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aids; motivational interviewing; counseling; rehabilitation
MeSH Terms: conditions — Hearing Loss | interventions — Standard of Care; Therapeutics; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-of-Care (Active Comparator): The "standard-of-care" control group will review and practice with the audiologist content such as: 1) information on hearing-aid batteries and how to change them, 2) cleaning/daily care of the hearing aids, and 3) inserting and removing the hearing aids.
  Interventions: Behavioral: Standard-of-Care
- Treatment (Experimental): The treatment group, on the other hand, will use a motivational tool (exploring importance) in a manner that is consistent with the spirit of motivational interviewing.
  Interventions: Behavioral: Treatment

INTERVENTIONS:
Behavioral: Standard-of-Care — the standard of care in audiologic practice
  Arms: Standard-of-Care
Behavioral: Treatment — motivational interviewing
  Other Names: Motivational Interviewing
  Arms: Treatment

SUMMARY:
The purpose of this study is to compare two different ways of helping first-time hearing-aid users get the most out of their hearing aids and determine if one method is better than the other. One method provides the patient with routine information regarding the care and use of hearing aids the other method uses tools to address patient-specific barriers against and motivators for hearing-aid use.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 20 and 89 years
* be a first-time hearing-aid user
* air-conduction pure-tone averages (mean thresholds at 500 Hz, 1000 Hz, and 2000 Hz) of 70 dB HL or less in both ears
* word-recognition scores of 40% or better in each ear
* English as their first language
* have sufficient vision and reading ability
* have the appropriate cognitive skills to participate in the study as determined by the Mini Mental State Exam, 2nd Edition - Brief Version (Folstein et al., 2010)
* have been fit by the VA Portland Health Care System Audiology and Speech Pathology Service (ASPS) with two hearing aids which have datalogging capabilities
* be independent in their completion of activities in daily living, as determined by their score on the Katz Index of Independence in Activities of Daily Living (Katz et al., 1970)
* have poor adoption of their hearing aids
* be free of a documented diagnosis in the VA Computerized Patient Record System (CPRS) record of neurological or psychological disorder, such as Alzheimer's disease, schizophrenia, or uncontrolled substance abuse, which would interfere with the completion of the study. Vulnerable populations are not being studied.

Exclusion Criteria:

Failure to satisfy any of the requirements listed as inclusion criteria

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Samantha Lewis, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz S, Downs TD, Cash HR, Grotz RC. Progress in development of the index of ADL. Gerontologist. 1970 Spring;10(1):20-30. doi: 10.1093/geront/10.1_part_1.20. No abstract available. PMID 5420677
- [Result] Cox RM, Stephens D, Kramer SE. Translations of the International Outcome inventory for Hearing Aids (IOI-HA). Int J Audiol. 2002 Jan;41(1):3-26. doi: 10.3109/14992020209101307. No abstract available. PMID 12467365

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects were consented but not enrolled into the study because they did not meet the inclusion criteria. One subject withdrew from the study after enrollment but prior to randomization.
Period: Overall Study
Arm/Group | Standard-of-Care | Treatment
Started | 11 (Number of participants randomized to standard-of-care.) | 10 (Number of participants randomized to treatment.)
Per Protocol Population | 11 | 9 (A subject was randomized to treatment but received standard of care and is not in the analyses.)
Completed | 10 (Final number of standard-of-care participants.) | 10 (Number of subjects who received the treatment that completed collection of outcome measures)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol population reported: One subject randomized to the "Treatment" erroneously received "Standard of Care" and is not included in this baseline report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-Care | Treatment | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Difference in Hours of Hearing Aid Use Between Pre-intervention and Post-intervention
Description: Hearing aid use was measured by the number of hours of use recorded in the hearing-aid software. This was measured on up to four occasions: Visit #1 to #3 (pre-intervention), and Visit #4 (post-intervention). Average daily hours of hearing aid use was documented at each time point, so that the Visit #4 observation is a measure of the average daily use between the start of intervention (Visit #3) and visit #4. Data logger results were averaged between the left and right hearing aids at each time point and across all three pre-intervention time points.
Time Frame: Collected pre-intervention and again at post-intervention appointment occurring between four and six weeks after the intervention date
Population: Standard-of-care group: one subject withdrew prior to the collection of outcome measures and one subject did not give valid data log measurement. These subjects are not included.
  Treatment: Three subjects did not give valid outcome data log measurement and one did not give a valid baseline measure. These subjects are not included.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard-of-Care | Treatment
Number analyzed (Participants) | 9 | 5
hours | -2.1 (3.3) | 2.2 (3.3)

2. Secondary Outcome: Difference Between Pre-intervention and Post-intervention Total Score on International Outcome Inventory for Hearing Aids
Description: The total score from the International Outcome Inventory for Hearing Aids (IOI-HA; Cox et al., 2000) was used to assess overall hearing-aid outcome. This measure consists of seven items assessing (1) daily hearing-aid use, (2) benefit, (3) residual activity limitation, (4) satisfaction, (5) residual participation restriction, (6) impact (of hearing impairment) on others, and (7) quality of Life. Responses to each question range from 1 (poorest) to 5 (best), for a total score range from 7 points to 35 points. The reported measurement was the change in total score from pre-intervention to post-intervention, with a maximum possible change of 28 points.
Time Frame: Collected twice once at pre-intervention visit and once at a post-intervention visit occurring four to six weeks following the intervention
Population: In the standard-of-care group, one subject withdrew from the study prior to the collection of outcome measures. In the treatment group, one subject did not answer one of the questions on the baseline questionnaire, thereby preventing calculation of a total score. This subject's data is therefore not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard-of-Care | Treatment
Number analyzed (Participants) | 10 | 8
units on a scale | 1.3 (2.9) | 0.4 (4.8)

ADVERSE EVENTS:
Time Frame: This was a minimal risk study. Adverse events were only monitored during study visits.
Arm/Group | Standard-of-Care | Treatment
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes